CLINICAL TRIAL: NCT03116165
Title: Cognitive-Behavioural Therapy as a Preventive Treatment for Post Traumatic Stress Disorder: An Randomized Controlled Trial in the Acute Trauma Care
Brief Title: Cognitive-Behavioural Therapy as a Preventive Treatment for Post Traumatic Stress Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisational changes in hospital which changed recruitment rates
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPN 2015/1820-31
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified prolonged exposure therapy (Experimental): Participants will receive three sessions of modified prolonged exposure therapy.
  Interventions: Behavioral: Modified prolonged exposure therapy
- Attention control (Placebo Comparator): Participants will receive three sessions of supportive counselling and psychoeducation
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Modified prolonged exposure therapy — Participants will receive three sessions of modified prolonged exposure therapy.
  Arms: Modified prolonged exposure therapy
Behavioral: Attention control — Participants will receive three sessions of supportive counselling and psychoeducation
  Arms: Attention control

SUMMARY:
This study will examine the use of modified prolonged exposure therapy in trauma patients recently exposed to trauma in an emergency room to prevent the onset of post-traumatic stress disorder.

DETAILED DESCRIPTION:
This study investigates if prolonged exposure is an effective treatment in reducing PTSD symptoms people who have recently experienced trauma. The study will also investigate predictive markers of PTSD, moderators of successful treatment and health economic aspects of the intervention.

Participants will first undergo an evaluation session that will include an interview (Immediate Stress Reaction Checklist) and questionnaires. Participants will subsequently be randomly assigned to receive either modified prolonged exposure therapy or attention control, starting the assigned intervention immediately. Participants in each arm will receive three weekly treatment sessions. Treatment will involve psychoeducation about common reactions to trauma, imaginal exposure (revisiting memories of a recent trauma out loud with a therapist and audio-recording these for review at home), exposure in vivo and breathing retraining. All participants will undergo assessments 2, 6 (primary endpoint) and 12 months after the intervention by blinded assessors. Patients unable to come to the clinic for follow-up assessments will be interviewed via telephone or skype. Source data will be quality monitored by an independent party (Karolinska trial alliance) according to the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the emergency department at the Karolinska University hospital Solna in the past 72 hours before the intervention
* Meets diagnostic criterion A for post-traumatic stress disorder in the fifth version of Diagnostic and Statistical Manual of Mental Disorders, DSM-5

Exclusion Criteria:

* Do not want to participate in the study
* Ongoing intoxication (e.g. severe alcohol intoxication)
* Other serious psychiatric comorbidity that demands attention (e.g. manic episode, acute suicidal ideation)
* Not oriented
* Not having a memory ot the tramatic event

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
CLINICIAN-ADMINISTERED PTSD SCALE for Diagnostic and Statistical Manual of Mental Disorders-5 (CAPS) | Change 2-, 6- (primary endpoint) and 12 months after intervention
  Clinical interview that gives a continuous measure of PTSD severity and dichotomous diagnosis of PTSD

SECONDARY OUTCOMES:
PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 (PCL-5) | Change 2-, 6- (primary endpoint) and 12 months after intervention
  Self-report questionnaire for the assessment of PTSD severity
Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) | Change from baseline to 2, 6 (primary endpoint) and 12 months after intervention
  Self-report questionnaire for the assessment of severity of depression
Euroqol (EQ-5D) | Measured 6 months after intervention
  Measure of general health and quality of life
WHO Disability Assessment Schedule (WHODAS) | Change 2-, 6- (primary endpoint) and 12 months after intervention
  Measure of general health and function
Adverse events | Change 2-, 6- (primary endpoint) and 12 months after intervention
  Measure of number adverse events
Subjective unit of distress scale (SUD) | Change at week 1, week 2 and week 3
  Ratings of distress
Intrusion diary | Change at week 1, week 2 and week 3
  A self-report diary on number of intrusions
Insomnia Severity Index (ISI) | Change 2-, 6- (primary endpoint) and 12 months after intervention
  Self-report questionnaire regarding insomnia
Multidimensional Scale of Perceived Social Support (MSPSS) | Change 2-, 6- (primary endpoint) and 12 months after intervention
  A measure to assess for social support
Trimbos Institute of costs in psychiatry (TIC-P) | Measured at 6 (primary endpoint) months after the intervention
  Self-report measure on societal costs

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden